CLINICAL TRIAL: NCT00756730
Title: Randomized, Open-label Study of Switch From Lopinavir/Ritonavir (LPV/r) or Fosamprenavir/Ritonavir (FPV/r) to Either Once Daily Atazanavir/Ritonavir (ATV/r) or Once Daily Darunavir/Ritonavir (DRV/r) (Plus Background Nucleoside Reverse Transcriptase Inhibitors) in Patients Experiencing Triglyceride Elevations While Receiving LPV/r or FPV/r.
Brief Title: Lopinavir/r or Fosamprenavir/r Switch to Atazanavir/r or Darunavir/r
Acronym: LARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-09
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections
Keywords: lopinavir; ritonavir; atazanavir; fosamprenavir; darunavir; anti-retroviral; AIDS; HIV; LARD; triglyceride; protease inhibitors; treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — atazanavir, ritonavir drug combination

ARMS (2):
- Switch to DRV/r (800mg/100mg) QD (Other): We designed a study to determine if switching virologically suppressed patients on a regimen containing LPV/r or FPV/r to either DRV/r or ATV/r would result in improved TGs while maintaining virological suppression. For this arm the sbject switched to DRV/r at a dose 800mg/100mg QD for 24 weeks. Subjects will continue to maintain their background NRTI drugs throughout the screening period and during the entire study.
  Interventions: Drug: DRV/r
- Switch to ATV/r (300mg/100mg QD) (Other): We designed a study to determine if switching virologically suppressed patients on a regimen containing LPV/r or FPV/r to either DRV/r or ATV/r would result in improved TGs while maintaining virological suppression. For this are the subject switched to ATV/r at a dose of 300mg/100mg QD for 24 weeks. Subjects will continue to maintain their background NRTI drugs throughout the screening period and during the entire study
  Interventions: Drug: ATV/r

INTERVENTIONS:
Drug: ATV/r — Switch to ATV/r at a dose of 300mg/100mg QD for 24 weeks. Subjects will continue to maintain their background NRTI drugs throughout the screening period and during the entire study.
  Other Names: Atazanavir/r
  Arms: Switch to ATV/r (300mg/100mg QD)
Drug: DRV/r — We designed a study to determine if switching virologically suppressed patients on a regimen containing LPV/r or FPV/r to either DRV/r or ATV/r would result in improved TGs while maintaining virological suppression. Switch to DRV/r at a dose 800mg/100mg QD for 24 weeks. Subjects will continue to maintain their background NRTI drugs throughout the screening period and during the entire study.
  Arms: Switch to DRV/r (800mg/100mg) QD

SUMMARY:
For participants with HIV taking either lopinavir or fosamprenavir who have elevated triglycerides, this trial will study the change in triglycerides after switching protease inhibitors.

DETAILED DESCRIPTION:
This Phase IV trial will look at lipid and virologic responses after a switch to a more lipid-friendly antiretroviral regimen. Participants will be randomized to receive either boosted atazanavir or boosted darunavir given once daily, along with background NRTIs. This 24-week study will require 4 visits after randomization for evaluation, monitoring, and lab studies.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving Antiretroviral Therapy (ART) regimen including LPV/r or FPV/r and > or equal to 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs). Patient must be on a stable regimen containing LPV/r or FPV/r for at least 12 weeks prior to screening.
* Documentation of an undetectable Human Immunodeficiency Virus (HIV) viral load (VL<400 copies/ml) using an FDA approved assay for a minimum of twelve weeks prior to screening AND undetectable HIV viral load using an FDA approved ultrasensitive assay at screening.
* No evidence of HIV protease resistance as defined by the Stanford HIV database
* Currently receiving first protease inhibitor unless switch to LPV/r or FPV/r was for non-virologic reasons
* Fasting triglycerides > 200 mg/dL
* No ongoing issues that in the opinion of the investigator would lead to decreased ability to comply with the study procedures
* If currently receiving a proton pump inhibitor, the dose is < omeprazole 20 mg or the equivalent dose of another proton pump inhibitor
* If patient is receiving another lipid lowering medication, it must be at a stable dose

Exclusion Criteria:

* Currently receiving an ART regimen other than > or equal to two NRTIs and either LPV/r or FPV/r
* Prior use of darunavir or atazanavir
* CDC Class C Illness diagnosed within 30 days of screening
* Patient is currently receiving the following Hydroxamethylglutaryl-coA (HMGCoA) reductase inhibitor medications (statins): pravastatin, lovastatin, simvastatin
* Patient is currently receiving a bile acid sequestrant (cholestyramine, colestipol, and colesevelam)
* Grade 3 or 4 Laboratory abnormalities as defined by a standardized grading scheme based on the DAIDS table with the following exceptions:

  1. Pre-existing diabetes mellitus with asymptomatic, nonfasting glucose grade 3 elevations
  2. Subjects with asymptomatic grade 3 fasting triglyceride or cholesterol elevations
* Clinical or laboratory evidence of clinically significant liver impairment/dysfunction disease or cirrhosis
* Note: Individuals co-infected with chronic hepatitis B or C viruses will be allowed to enter the trial if their condition is clinically stable and they will not require therapy during the course of the study. Individuals diagnosed with acute viral hepatitis at screening will not be allowed to enroll during acute phase
* Active substance abuse or significant psychiatric illness that in the opinion of the investigator might interfere with study compliance
* Use of any investigational agents 30 days prior to screening
* Life expectancy < 6 months in the opinion of the investigator
* Pregnancy or breast feeding
* Female subject of childbearing potential (i.e., heterosexually active, and not surgically sterile or at least two years post-menopausal) not using effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last trial related activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Skiest, MD, Principal Investigator — Community Research Initiative
Locations (11):
- United States (11):
  - Spectrum Medical Group, Phoenix, Arizona
  - AIDS Healthcare Foundation, Los Angeles, California
  - Orlando Immunology Center, Orlando, Florida
  - Community Research Initiative, Boston, Massachusetts
  - Community Research Initiative - West, Springfield, Massachusetts
  - Abbott Northwestern Infectious Disease and Travel Clinic, Minneapolis, Minnesota
  - AIDS Community Health Center, Rochester, New York
  - Philadelphia Fight, Philadelphia, Pennsylvania
  - David M. Lee, M.D., P.A., a/b/a Uptown Physicians Group, Dallas, Texas
  - Nicholaos C. Bellos, MD, PA, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD: Virologically suppressed patients on a regimen containing Lopinavir/ritonavir (LPV/r) or fosamprenavir/ritonavir (FPV/r) were switched to DRV/r, 800mg/100mg QD
- Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD: Virologically suppressed patients on a regimen containing Lopinavir/ritonavir (LPV/r) or fosamprenavir/ritonavir (FPV/r) were switched to ATV/r
Period: Overall Study
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Started | 25 | 24
Completed | 25 | 22
Not Completed | 0 | 2
Not completed — discontinued due to rash prior to week 4 | 0 | 1
Not completed — persistent low-level viremmia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Customized [Mean (Full Range); unit: years] | 48 [34 to 67] | 46 [30 to 60] | 47 [30 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 19
  Not Hispanic or Latino | 18 | 11 | 29
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49
CD4 Count [Mean (Full Range); unit: cells/mm3] | 584 [249 to 996] | 554 [31 to 1066] | 569 [31 to 1066]
Viral Load [Number; unit: copies/mL] | NA [NA to NA] — VL was not detected. All values were reported less than 50 copies/ml, the lower limit of detection. | NA [NA to NA] — VL was not detected. All values were reported less than 50 copies/ml, the lower limit of detection. | 0 [NA to NA]
Baseline antiretroviral medications - Protease inhibitors [Number; unit: participants]
  Lopinavir/ritonavir (LPV/r) | 23 | 23 | 46
  fosamprenavir/ritonavir (FPV/r) | 2 | 1 | 3
Baseline medications - Nucleoside analogs [Number; unit: Participants]
  viread (TDF)/emtriva (FTC) | 15 | 17 | 32
  ziagen (ABC)/Epivir (3TC) | 5 | 5 | 10
  other | 5 | 2 | 7
Lipid Lowering Medications [Number; unit: participants]
  statin | 6 | 3 | 9
  fibrate | 5 | 6 | 11
  fish oil | 5 | 3 | 8
  niacin | 0 | 1 | 1
  none | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Experience 10% Decline in Triglycerides From Baseline to Week 24.
Description: A 10% decline in triglycerides (TGs) was determined to be clinically significant. The percentage of people that experienced a 10% decline was calculated by dividing the number who had a decline of 10% TGs by the total number of participants in the arm.
Time Frame: baseline, 24 weeks
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia. Neither subject met criteria for virologic failure.
Measure: Number; unit: percentage of patients
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
percentage of patients | 80 | 73

2. Secondary Outcome: Percent of Patients With HIV VL <200 Copies/mL at Week 4, 12 & 24
Time Frame: Week 4, 12 & 24
Measure: Number; unit: percentage of participants
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 24
percentage of participants
  Week 4 | 100 | 100
  Week 12 | 100 | 100
  Week 24 | 100 | 100

3. Secondary Outcome: Difference in CD4 From Baseline to Week 24
Time Frame: baseline to Week 24
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
cells/mm^3 | 10.75 (17.67) | 14.28 (19.77)

4. Secondary Outcome: Total Cholesterol in the Two Study Groups at 24 Weeks
Time Frame: Week 24
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
mg/dL | 195 [110 to 311] | 195 [132 to 304]

5. Secondary Outcome: LDL Cholesterol at Week 24
Time Frame: week 24
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
mg/dL | 116 [55 to 180] | 111 [46 to 204]

6. Secondary Outcome: HDL Cholesterol at Week 24
Time Frame: 24 weeks
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
mg/dL | 38 [22 to 54] | 40 [26 to 55]

7. Primary Outcome: At Week 24 the Percentage of Subjects That Had Triglycerides Less Than 200 mg/dL
Time Frame: 24 weeks
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Number; unit: percentage of participants
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
percentage of participants | 48 | 55

8. Primary Outcome: The Change in Fasting Triglyceride Level From Baseline to Week 24
Time Frame: Baseline to week 24
Population: Two patients in the ATV/r arm discontinued prior to week 24: 1 due to a grade 2 rash, and one due to low level viremia.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Number analyzed (Participants) | 25 | 22
mg/dL | -126 [-312 to 133] | -88 [-469 to 90]

ADVERSE EVENTS:
Time Frame: Baseline to 24 weeks
Arm/Group | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/24
Other Adverse Events (participants affected / at risk) | 7/25 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD (N=25) | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD (N=24)
possible bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
alcohol withdrawal/suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
urosepsis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch to Darunavir/Ritonavir (DRV/r) , 800mg/100mg QD (N=25) | Switch to Atazanavir/Ritonavir (ATV/r), 300mg/100mg QD (N=24)
Upper Respiratory Infection (URI) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erectile Dysfunction (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes